CLINICAL TRIAL: NCT00005508
Title: Determinants of Coronary Disease in High Risk Families
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5026; R01HL059684 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To define factors contributing to coronary heart disease (CHD) in high risk families.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study followed healthy siblings of patients diagnosed with CHD before age 60. All siblings underwent comprehensive risk factor screening and exercise thallium tomography to identify occult CHD. Follow-up was performed from 6-15 years after entry (mean 8.7 years) to determine the incidence of (1) acute coronary events (sudden death, myocardial infarction, and unstable angina) and (2) progression of occult CHD (repeat exercise thallium tomography). Blood was obtained for genomic DNA, which was tested for polymorphisms of candidate genes which may be associated with premature thrombotic CHD events (platelet proteins GPIIB/IIIa[PlA1/A2 and Baka/b] and GPIbB, endothelial nitric oxide synthase, angiotensin converting enzyme, angiotensinogen, D-fibrinogen, plasminogen activator-1, and methylenetetrahydrofolate reductase). Plasma levels of proteins implicated in the pathogenesis of atherosclerosis and thrombotic CHD events were measured (fibrinogen, plasminogen activator inhibitor-1, tissue plasminogen activator, homocysteine, lipoprotein (a), and apo(a) isoform size). DNA was also obtained from living probands and affected siblings to use for genetic linkage studies using affected and unaffectedsibling pairs. Statistical analyses examined (1) whether selected genetic polymorphisms were linked to the occurrence of acute CHD events, and (2) to what extent traditional sociodemographic and biological coronary risk factors or new genetic polymorphisms explained the progression of occult CHD, or the transition from occult to symptomatic CHD events in families with premature CHD.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Becker — Johns Hopkins University